CLINICAL TRIAL: NCT05614466
Title: SIMPLY-B Study - A Pilot Evaluation of a Primary Care E-support Package of Automated Case Finding, Simplified Treatment Algorithm and Decision Support to Increase Hepatitis B Treatment Uptake in Primary Care Clinics
Brief Title: The SIMPLY-B Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nadine Barnes (Other)
Responsible Party: Sponsor-Investigator, Nadine Barnes, Manager, Research Grants and Research Integrity Office, Macfarlane Burnet Institute for Medical Research and Public Health Ltd
Organization: Macfarlane Burnet Institute for Medical Research and Public Health Ltd (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SIMPLY-B Study
Record Dates: First submitted 2022-10-25; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Hepatitis B Virus Related Hepatocellular Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients living with hepatitis B (Experimental): Patients living with hepatitis B will be managed at the GP clinic using the Simply B e-support package
  Interventions: Other: The Simply B Study

INTERVENTIONS:
Other: The Simply B Study — This study will be conducted in three parts:
  Part A: A prospective open label pilot intervention study, comparing the proportion of people with hepatitis B who are managed by their GP in primary care clinics before, 12 months and 24 months after implementation of the Simply B electronic hepatitis B support package.
  Part B: A nested qualitative health services feasibility study using semi -structured interviews and thematic analysis Part C: A mathematical modelling study using a Markov model to determine cost effectiveness of Simply B for increasing hepatitis B treatment uptake compared to status quo of hospital care.

SUMMARY:
This study will be conducted in three parts:

Part A: A prospective open label pilot intervention study, comparing the proportion of people with hepatitis B who are managed by their GP in primary care settings before, 12 months and 24 months after implementation of the Simply B electronic hepatitis B support package.

Part B: A nested qualitative health services feasibility study using semi -structured interviews and thematic analysis

DETAILED DESCRIPTION:
The Simply B electronic GP support package consists of:

1. Semi-automated hepatitis B case-finding in the primary care clinic using clinic EMR software
2. Automated blood test ordering using clinic EMR software
3. A simplified hepatitis B treatment algorithm and online e-support tool that provides the GP with a simplified management plan based on clinical data entered into the tool by generating a hepatitis B chronic disease management plan.
4. Automated rapid linkage to specialist support through the e-support tool, with a follow up call from a specialist nurse provided within two business days of the initial patient/GP consultation.
5. Clinical data collection through the e-support tool into an online secure database, visible by the GP and hospital specialist, allowing automated reminders and monitoring of timely and appropriate hepatitis B management steps.
6. Linkage of de-identified data drawn from the Simply B database to the ACCESS and PATRON surveillance network to allow monitoring of progress toward National Strategy Hepatitis B treatment targets in primary care.

The e-support tool is based on an online RedCAP database accessible to both the GP and St Vincent's hospital specialist team via different interfaces and stored securely on the St Vincent's Hospital Cloud. The investigators have partnered with the Future Health Today (FHT) software development team (University of Melbourne) to integrate the Simply B e-support package into primary care electronic medical record software.

The GP enters demographic and pathology result data into a simple online data entry form. Based on a simplified hepatitis B management algorithm, this determines treatment eligibility and immediately generates an automatic patient management plan. For clinics that are part of the FHT network, FHT extracts demographic and pathology result data automatically and populates the Simply B tool, therefore the GP does not need to manually enter any data. Instructions of how to treat, monitor and perform liver cancer surveillance are included in the automated management plan.

The hospital specialist nurse and specialist clinicians have online access to the 'back end' of the Simply B e-support tool database, allowing them to monitor and enter data. This database contains all the demographic and clinical data entered by the GP in the e-support tool data entry form and automatically generates dates for follow up review, including date of next liver cancer surveillance if the patient fulfils eligibility criteria. Upcoming milestone appointments trigger alert emails to the GP and specialist hepatitis nurses facilitating timely hepatitis B management.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years
2. Attended participating primary care clinic in the preceding 36 months (June 1, 2019-June 30, 2022) or attended the clinic during the study period
3. HBsAg positive
4. Treatment naïve
5. Not receiving specialist hepatitis B care

Exclusion Criteria:

1. < 18 years of age
2. Already on hepatitis B treatment
3. Already attending hepatitis B specialist care
4. Hepatitis C or hepatitis D coinfection
5. HIV coinfection
6. Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients previously diagnosed with chronic hepatitis B within each primary care clinic study site who have attended the clinic within the 36-month period prior to implementation of the intervention | 36 months prior to study
  Number of patients previously diagnosed with chronic hepatitis B within each primary care clinic study site who have attended the clinic within the 36-month period prior to implementation of the intervention
Number (proportion) of hepatitis B patients receiving guideline-based hepatitis B management by GP | 2 years
  Number (proportion) of hepatitis B patients receiving guideline-based hepatitis B management by GP
Number (proportion) of hepatitis B patients receiving specialist care in a hospital or private setting | 2 years
  Number (proportion) of hepatitis B patients receiving specialist care in a hospital or private setting
Number (proportion) of hepatitis B patients receiving treatment by the GP in primary care | 2 years
  Number (proportion) of hepatitis B patients receiving treatment by the GP in primary care

SECONDARY OUTCOMES:
Acceptability and feasibility of using the Simply B package to facilitate hepatitis B management by GPs in primary care from health worker and patient perspectives. | 2 years
  Acceptability and feasibility of using the Simply B package to facilitate hepatitis B management by GPs in primary care from health worker and patient perspectives. This will be done via a 12-month post implementation semi-structured interview with GPs, nurses, practices managers and patients living with hepatitis B.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moussa D, Wallace J, Manski-Nankervis JA, Doyle JS, Nguyen L, Boyle D, Stoove MA, Asselin J, Valaydon Z, Ahad M, Glasgow S, New K, Hocking JS, Sanci L, Thompson A, Hellard M, Howell J. Assessment of a primary care e-support package of automated case finding, simplified treatment algorithm and decision support to increase hepatitis B treatment uptake in primary care clinics in Australia (SIMPLY-B Study): protocol for a pilot evaluation. BMJ Open. 2023 Mar 16;13(3):e070663. doi: 10.1136/bmjopen-2022-070663. PMID 36927591